CLINICAL TRIAL: NCT05825950
Title: Predicting Outcomes in Intermediate and High-risk Non-muscle Invasive Bladder Cancer Using Automated Analysis of Digital Pathology Data
Brief Title: Artificial Intelligence Prediction Tool in Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Valar Labs (Unknown)
Responsible Party: Principal Investigator, Solomon Woldu, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-0188
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: NMIBC; Bladder cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HR NMIBC group: High Risk (HR) NMIBC group of participants studied include ones with American Urological Association (AUA) / Society of Urologic Oncology (SUO) criteria such as : high grade T1, recurrent high grade Ta, high grade Ta >3 cm, multifocal high grade Ta, any Carcinoma in-situ (CIS), any BCG failure in high grade disease, any variant histology, any lymphovascular invasion.
  Note: Ta means the cancer is just in the innermost layer of the bladder lining. T1 means the cancer has started to grow into the connective tissue beneath the bladder lining.
- IR NMIBC group: Intermediate Risk (IR) NMIBC group of participants studied include ones with AUA/SUO criteria such as : recurrence within 1 year low grade Ta, solitary low grade Ta >3 cm, multifocal low grade Ta, high grade Ta ≤3 cm, low grade T1 Note: Ta means the cancer is just in the innermost layer of the bladder lining. T1 means the cancer has started to grow into the connective tissue beneath the bladder lining.

SUMMARY:
This is a multi-center study and the aim is to develop and validate an Artificial Intelligence (AI) -based histologic analysis tool to predict responsiveness to intravesical Bacillus Calmette-Guérin (BCG) and intravesical chemotherapy in intermediate and high-risk non-muscle invasive bladder cancer patients.

DETAILED DESCRIPTION:
Analysis will be performed on the most recent Transurethral resection of bladder tumor (TURBT) histologic specimen obtained prior to BCG induction and on histologic specimens at time of recurrence after BCG induction. This stratification is of potential utility to clinicians for patient counseling purposes, for the identification of patients likely to benefit from induction or re-induction with BCG, and for consideration of alternative treatment strategies including clinical trials, chemotherapy, or cystectomy. Additionally, there is currently no reliable tool for identifying which NMIBC patients are most likely to benefit from adjuvant BCG versus intravesical chemotherapy. This is of current relevance in the management of Intermediate-risk (IR) NMIBC since both BCG and chemotherapy are first-line treatment options and will likely become of increasing relevance in High-risk (HR) NMIBC as efficacious first-line alternatives to intravesical BCG are introduced into clinical practice. In the proposed prospective study, the study team also aims to develop and then validate an AI-based histologic analysis tool for clinicians that is intended to predict recurrence following intravesical chemotherapy in IR and HR NMIBC patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intermediate or high-risk non-muscle invasive bladder cancer as defined by AUA/SUO criteria (Intermediate-risk: recurrence within 1 year low grade Ta, solitary low grade Ta >3 cm, multifocal low grade Ta, high grade Ta ≤3 cm, low grade T1; High risk: high grade T1, recurrent high grade Ta, high grade Ta >3 cm, multifocal high grade Ta, any CIS, any BCG failure in high grade disease, any variant histology, any lymphovascular invasion) following pathologic evaluation of tissue specimens from TURBT.
* Intravesical therapy within 6 months from enrollment including patients treated with BCG, mitomycin C, or Gemcitabine/Docetaxel.
* English or Spanish speakers
* ≥ 18 years of age
* Ability to understand and the willingness to provide an informed consent

Exclusion Criteria:

* Inadequate tissue from TURBT
* ≥ T2 bladder cancer
* Systemic therapy
* Inability to read or write English or Spanish
* Unwilling to sign written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified in urology clinics after a diagnosis of non-muscle invasive bladder cancer undergoing intravesical BCG therapy or chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) at 3 months after TURBT in participants with HR NMIBC | 3 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of first procedure confirming histopathological recurrence, disease progression or death as a first event from any cause during surveillance cystoscopy at 3 months.
Recurrence free survival (RFS) at 6 months after TURBT in patients with HR NMIBC | 6 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of first procedure confirming histopathological recurrence, disease progression or death as a first event from any cause during surveillance cystoscopy at 6 months.
Recurrence free survival (RFS) at 12 months after TURBT in patients with HR NMIBC | 12 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of first procedure confirming histopathological recurrence, disease progression or death as a first event from any cause during surveillance cystoscopy at 12 months.
Recurrence free survival (RFS) at 24 months after TURBT in patients with HR NMIBC | 24 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of first procedure confirming histopathological recurrence, disease progression or death as a first event from any cause during surveillance cystoscopy at 24 months.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) at 3 months following the first negative surveillance cystoscopy after TURBT in patients with IR NMIBC | 3 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of negative surveillance cystoscopy after TURBT confirming histopathological recurrence, disease progression or death as a first event from any cause at 3 months.
Recurrence free survival (RFS) at 6 months following the first negative surveillance cystoscopy after TURBT in patients with IR NMIBC | 6 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of negative surveillance cystoscopy after TURBT confirming histopathological recurrence, disease progression or death as a first event from any cause at 6 months.
Recurrence free survival (RFS) at 12 months following the first negative surveillance cystoscopy after TURBT in patients with IR NMIBC | 12 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of negative surveillance cystoscopy after TURBT confirming histopathological recurrence, disease progression or death as a first event from any cause at 12 months.
Recurrence free survival (RFS) at 24 months following the first negative surveillance cystoscopy after TURBT in patients with IR NMIBC | 24 months
  Recurrence free survival (RFS) is measured as the time from start of clinical treatment / study enrollment to the date of negative surveillance cystoscopy after TURBT confirming histopathological recurrence, disease progression or death as a first event from any cause at 24 months.
Progression-free survival (PFS) at 12 months following the first negative surveillance cystoscopy after TURBT in patients with HR or IR NMIBC | 12 months
  Progression-Free Survival is measured as the time from the patient registration to the date of first negative surveillance cystoscopy after TURBT in patients with HR or IR NMIBC or death from any cause in the absence of progression, whichever occurs first. An increase in tumor stage and/or the presence of muscle invasive disease diagnosed during surveillance cystoscopy will constitute disease progression.
Progression-free survival (PFS) at 24 months following the first negative surveillance cystoscopy after TURBT in patients with HR NMIBC or IR NMIBC | 24 months
  Progression-Free Survival is measured as the time from the patient registration to the date of first negative surveillance cystoscopy after TURBT in patients with HR or IR NMIBC or death from any cause in the absence of progression, whichever occurs first. An increase in tumor stage and/or the presence of muscle invasive disease diagnosed during surveillance cystoscopy will constitute disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No